CLINICAL TRIAL: NCT04990427
Title: A Phase 1 Open-Label, Proof-of-Concept Study to Evaluate the Safety and Efficacy of CLBS201 Autologous Peripheral Blood-Derived CD34+ Cells in Subjects with Chronic Kidney Disease and Type 2 Diabetes Mellitus
Brief Title: CLBS201 in Patients with Chronic Kidney Disease (CKD) and Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLBS201-P01a
Record Dates: First submitted 2021-07-30; First posted 2021-08-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney disease; Type 2 Diabetes Mellitus; Diabetic Kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLBS201 (Experimental): CLBS201 will be administered in an open-label fashion via intra-renal-arterial infusion in 6 subjects followed by 6 months of observation.
  Interventions: Drug: CLBS201

INTERVENTIONS:
Drug: CLBS201 — 1 x 10^6 to 300 x 10^6 autologous CD34+ cells

SUMMARY:
CLBS201 will evaluate the safety, tolerability, and therapeutic effect in subjects with CKD and T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 75 years, inclusive
2. Documented diagnosis of type 2 diabetes
3. eGFR of 30 to <45 mL/min/1.73m at the screening visit.
4. UACR 300 mg/g to ≤ 5000 mg/g

Exclusion Criteria:

1. Hemoglobin < 10 g/dL
2. Hemoglobin A1c ≥8% at the time of screening
3. Acute kidney injury within 6 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | 6 Months
  Proportion of patients with a treatment-emergent serious adverse event

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) | 6 Months
  Change in eGFR from baseline
UACR & UPCR | 6 Months
  Change in UACR & UPCR from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Buck, MD, Study Director — Lisata Therapeutics, Inc.
Locations (1):
- Clinical Advancement Center, PLLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No